CLINICAL TRIAL: NCT07230405
Title: A Phase II Study to Evaluate the Safety and Efficacy of SKB571 in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Phase II Study of SKB571 in Patients With Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB571-II-02
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer (Non-Small Cell)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB571 monotherapy (Experimental)
  Interventions: Drug: SKB571 for injection

INTERVENTIONS:
Drug: SKB571 for injection — SKB571 for injection is administered every 3 weeks(Q3W) until radiographic disease progression,intolerable toxicity, or other protocol-specified treatment discontinuation criteria, whichever occurs first.

SUMMARY:
This is a multicenter, phase II study. The purpose of this study is to evaluate the safety and preliminary anti-tumor activity of SKB571 in patients with advanced non-small cell lung cancer. Eligible subjects will receive SKB571 monotherapy, until radiographic disease progression, intolerable toxicity, discontinuation of study treatment required by the subject, or other protocol-specified treatment discontinuation criteria, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-75 years at the time of signing the informed consent form
2. Subjects with histologically or cytologically confirmed locally advanced or metastatic NSCLC .
3. Subjects with at least one measurable lesion assessed by the investigator according to RECIST v1.1.
4. Subjects with Eastern Cooperative Oncology Group (ECOG) status score of 0 or 1.
5. Subjects who are assessed by the investigator to have an expected survival of ≥ 12 weeks.
6. Subjects who have adequate organ function.
7. Subjects who have recovered from all toxicities due to prior therapy .
8. Male and female subjects must agree to use highly effective contraception methods during the study treatment.
9. Subjects who voluntarily sign the informed consent form.

Exclusion Criteria:

1. Subjects with known active or untreated central nervous system (CNS) metastases.
2. Subjects with other malignant tumors within 3 years prior to the first dose.
3. Subjects with history of major cardiovascular, cerebrovascular, or thromboembolic disease.
4. Subjects with human immunodeficiency virus (HIV) infection, or any known active viral hepatitis, or hepatitis B or hepatitis C.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites effusion requiring repeated drainage.
6. Subjects with known allergy or hypersensitivity to SKB571 or its excipients.
7. Subjects with clinically severe lung injuries due to pulmonary complications.
8. History of noninfectious pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
9. Subjects with major surgery within 28 days prior to the first dose.
10. Subjects who have received live vaccines within 30 days prior to the first dose of study treatment, or who are scheduled to receive live vaccines during the study.
11. Subjects who have received strong cytochrome P450 (CYP3A4) inhibitors or inducers, or BCRP inhibitors within 2 weeks prior to the first dose of study treatment or within 5 half-lives of known drug, whichever is longer.
12. Subjects who have received chemotherapy, immunotherapy, or biological therapy within 4 weeks prior to the first dose of study treatment.
13. Subjects with active infection requiring systemic anti-infective therapy within 14 days prior to the first dose of study treatment.
14. Subjects with any disease requiring systemic treatment with corticosteroids (prednisone at doses > 10 mg/d or similar drugs with equivalent doses) or other immunosuppressive therapy within 14 days prior to the first dose of study treatment.
15. Any condition that, in the opinion of the investigator, will interfere with the assessment of study treatment or the safety of the subject or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2028-01-19 (Estimated); Study Completion 2028-01-19 (Estimated)

PRIMARY OUTCOMES:
AE | Up to 24 months
  Incidence and severity of adverse events (AEs)
ORR | Up to 24 months
  Objective response rate (ORR) (assessed by the investigators as per RECIST v1.1)

SECONDARY OUTCOMES:
PFS | Up to 24 months
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
DOR | Up to 24 months
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
OS | Up to 24 months
  Time from start of treatment to death due to any reason.
DCR | Up to 24 months
  Disease control rate (DCR) (assessed by the investigators as per RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Henan Cancer Hospital, Zhengzhou